CLINICAL TRIAL: NCT00858182
Title: Evaluation of a New Peritoneal Dialysis Solutions Containing Glucose, Xylitol and L-carnitine Compared to Standard PD Solutions in End-stage Renal Disease (ESRD) Patients on Continuous Ambulatory Peritoneal Dialysis (CAPD)
Brief Title: Study of Safety and Efficacy on New Peritoneal Dialysis Solutions
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-001-07
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2013-03

CONDITIONS: End-Stage Renal Disease
Keywords: L-Carnitine; Xylitol; Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: PD solution for nocturnal exchanges
- Group B (Experimental)
  Interventions: Drug: PD solution for diurnal exchanges

INTERVENTIONS:
Drug: PD solution for nocturnal exchanges — Instillation of a PD solution containing xylitol (1.5%), L-carnitine (0.1%) and glucose (0.5%) for the nocturnal exchange in CAPD treated patients. PD solutions are instilled for 4 weeks.
  Arms: Group A
Drug: PD solution for diurnal exchanges — Instillation of a PD solution containing xylitol (0.6%), L-carnitine (0.1%) and glucose (0.5%) for the diurnal exchanges in CAPD treated patients. PD solutions are instilled for 4 weeks.
  Arms: Group B

SUMMARY:
A major challenge of peritoneal dialysis (PD) therapy is the development of glucose-sparing strategies able to provide an efficacious ultrafiltration (UF) profile. Study hypothesis is to evaluate the possibility to formulate PD solutions containing xylitol and L-carnitine as osmotic agents to partially replace glucose.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosis of ESRD treated for at least three month with CAPD, as stated by the medical staff of the center;
* CAPD treatment with 2.27% of glucose solution for the nocturnal exchange;
* Stable clinical condition within four weeks before screening period, certified by medical/surgical history, physical examination and laboratory exploration;
* Hemoglobin level ≥9g/dL;
* Residual diuresis ≤800mL;
* Absence of acute peritonitis and/or peritoneal catheter infection (either exit site or subcutaneous tunnel) episodes within three months before selection;
* Stable peritoneal permeability, as confirmed by a PET between 0.50 and 0.81 during previous three months and at day 0 of the screening period;
* Total urea Kt/V >1.5 per week at a control during previous three months and at day 0 of the screening period and/or minimal total creatinine clearance of 45 liter/week at a control during previous three months and at day 0 of the screening period; 1- To understand and sign an informed consent form.

For patients who will be included in Group B, the following criteria must be fulfilled too:

* Be treated with Extraneal (nocturnal exchange bag solution) for at least 1 month
* Be treated with 2 or 3 diurnal exchange bag solutions (solution bags with 1.36% or 2.27% glucose) and one nocturnal exchange bag solution (Extraneal)

Exclusion Criteria:

* History of alcohol or drug abuse in the last six months before selection for the study;
* Androgen therapy in the last six months before selection;
* Active infections;
* History of congestive heart failure stage III and IV NYHA;
* History of major cardiovascular events like stroke, acute myocardial infarction, coronary or other arterial revascularization procedures in the last three months before selection;
* Clinically relevant cardiac arrhythmia;
* Clinically relevant abnormalities of functional hepatic tests;
* Therapy with L-carnitine or its derivatives in the last three months before selection;
* Pregnancy, lactating women or female subjects of childbearing potential who do not use an effective method of contraception;
* Presence of relevant chronic medical conditions that could suggest exclusion of patient from the study or could interfere with assessment of study parameters, especially if the life expectation is less then one year;
* Participation in another clinical study within the past month;
* Known or supposed allergic reactions to L-carnitine or xylitol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2012-10 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
To assess ultrafiltration efficacy of PD solutions containing L-Carnitine and Xylitol | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Capusa, PhD, Study Director — "Dr Carol Davila" University Hospital of Nephrology, Romania; Gabriel Mircescu, PhD, Study Chair — "Dr Carol Davila" University Hospital of Nephrology, Romania